CLINICAL TRIAL: NCT02261493
Title: Evaluation of the Safety and Efficacy of Treatment With BOTOX® (Botulinum Toxin Type A) Purified Neurotoxin Complex for Subjects With Facial Rhytides (Forehead Lines, Glabellar Lines, Lateral Canthal Lines)
Brief Title: A Safety and Efficacy Study of OnabotulinumtoxinA in Upper Facial Rhytides
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 191622-143; 2014-001815-38 (EudraCT Number)
Record Dates: First submitted 2014-10-03; First posted 2014-10-10 (Estimated); Results first posted 2017-07-25 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-06

CONDITIONS: Facial Rhytides; Glabellar Rhytides
MeSH Terms: interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- OnabotulinumtoxinA Dose A (Experimental): OnabotulinumtoxinA Dose A injected into the protocol-specified areas on Day 1. Subjects will receive at least 1 and up to 3 treatments.
  Interventions: Biological: OnabotulinumtoxinA
- OnabotulinumtoxinA Dose B (Experimental): OnabotulinumtoxinA Dose B injected into the protocol-specified areas on Day 1. Subjects will receive at least 1 and up to 3 treatments.
  Interventions: Biological: OnabotulinumtoxinA
- Placebo followed by OnabotulinumtoxinA Dose A (Placebo Comparator): Placebo (normal saline) injected into the protocol-specified areas on Day 1. If the subject meets the re-treatment criteria, the subject will receive up to 2 treatments with onabotulinumtoxinA Dose A into the protocol-specified areas.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Biological: OnabotulinumtoxinA — OnabotulinumtoxinA injected into the protocol-specified areas. Subjects will receive at least 1 and up to 3 treatments.
  Other Names: BOTOX® Cosmetic; botulinum toxin Type A
  Arms: OnabotulinumtoxinA Dose A; OnabotulinumtoxinA Dose B
Drug: Normal Saline — Placebo (normal saline) injected into the protocol-specified areas on Day 1.
  Arms: Placebo followed by OnabotulinumtoxinA Dose A

SUMMARY:
This is a safety and efficacy study of onabotulinumtoxinA in subjects with upper facial rhytides (forehead lines, glabellar lines, lateral canthal lines [crow's feet lines]).

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe forehead lines, glabellar lines, and crow's feet lines
* Willing to have facial photos taken

Exclusion Criteria:

* Prior exposure to botulinum toxin of any serotype for any indication
* Anticipated need for treatment with botulinum toxin of any serotype for any indication during the study, other than study treatment
* Diagnosis of myasthenia gravis, Eaton-Lambert syndrome, or amyotrophic lateral sclerosis
* Any facial resurfacing laser or light treatment, microdermabrasion, or superficial peels in the past 3 months
* Any medium depth or deep depth facial chemical peels; facial skin resurfacing; or permanent facial make-up in the past 6 months
* Any nonpermanent soft tissue fillers, or treatment with oral retinoids in the past year - Prior face lift, thread lift, eyebrow lift, or related procedures (eg, eyelid and/or eyebrow surgery)
* Prior facial treatment with permanent soft tissue fillers, synthetic implants (eg, Gore-Tex®), and/or fat transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 787 (Actual)
Dates: Start 2014-10-27 (Actual); Primary Completion 2015-06-03 (Actual); Study Completion 2016-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (24):
- United States (10):
  - The Petrus Center for Aesthetic, Little Rock, Arkansas
  - Westside Aesthetics, Los Angeles, California
  - Eye Research Foundation, Newport Beach, California
  - Steve Yoelin, MD Medical Associates, Inc., Newport Beach, California
  - Baumann Cosmetic & Research Institute, Miami, Florida
  - Saint Louis University, St Louis, Missouri
  - The Center For Dermatology Cosmetic and Laser Surgery, Mount Kisco, New York
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - The Center for Skin Research, Houston, Texas
  - Premier Clinical Research, Spokane, Washington
- Belgium (3):
  - Aalst Dermatology Clinic, Aalst
  - UZ Brussel, Jette
  - Medical Skin Care - Sint-Truiden, Limbourg
- Germany (6):
  - Rosenpark Research, Darmstadt
  - Hautzentrum Koeln (Cologne Dermatology), Köln Nordrhein-Westfalen
  - Hautok und hautok-cosmetics, München
  - Praxisgemeinschaft Theatiner46, München
  - Hautzentrum am Starnberger See GmbH, Starnberg
  - CentroDerm Study Center, Wuppertal
- United Kingdom (5):
  - Shakespeare House Health Centre, General Practice, Basingstoke
  - Medizen Clinic, Birmingham
  - The Bosham Clinic, Chichester
  - Waverlery Medical Practice, Coatbridge
  - The Gatehouse, Whitegate

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were randomized to placebo, onabotulinumtoxinA Dose A, or onabotulinumtoxinA Dose B in Period 1. Subjects randomized to receive placebo or Dose B in Period 1, who subsequently continued to Period 2, received onabotulinumtoxinA Dose A in Period 2.
Groups:
- Placebo (Normal Saline) Followed by OnabotulinumtoxinA Dose A: Placebo (normal saline) injected into the protocol-specified areas on Day 1. If the subject meets the re-treatment criteria, the subject will receive up to 2 treatments with onabotulinumtoxinA Dose A into the protocol-specified areas.
Period: Overall Study
Arm/Group | Placebo (Normal Saline) Followed by OnabotulinumtoxinA Dose A | OnabotulinumtoxinA Dose B | OnabotulinumtoxinA Dose A
Started | 156 | 318 | 313
Completed | 126 | 271 | 287
Not Completed | 30 | 47 | 26
Not completed — Noncompliance | 0 | 0 | 2
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Undisclosed alcohol abuse | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Personal Reasons | 14 | 14 | 16
Not completed — Lost to Follow-up | 14 | 27 | 8
Not completed — Pregnancy | 1 | 2 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Normal Saline) Followed by OnabotulinumtoxinA Dose A | OnabotulinumtoxinA Dose B | OnabotulinumtoxinA Dose A | Total
Number analyzed (Participants) | 156 | 318 | 313 | 787
Age, Customized [Number; unit: Participants]
  <65 years | 147 | 300 | 302 | 749
  >=65 years | 9 | 18 | 11 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 278 | 284 | 702
  Male | 16 | 40 | 29 | 85

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With ≥2-Grade Improvement From Baseline on Both the Investigator's and Subject's Facial Wrinkle Scale (FWS) Ratings of Forehead Line Severity at Maximum Eyebrow Elevation
Description: The Investigator and subject each assessed the severity of the subject's forehead lines at maximum eyebrow elevation using the 4-grade FWS, where 0=none, 1=mild, 2=moderate, and 3=severe. The percentage of subjects with at least a 2-grade improvement from baseline assessed by both the Investigator and the subject are reported.
Time Frame: Baseline, Day 30
Population: Intent-to-Treat: all randomized subjects
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | Placebo (Normal Saline) Followed by OnabotulinumtoxinA Dose A | OnabotulinumtoxinA Dose B | OnabotulinumtoxinA Dose A
Number analyzed (Participants) | 156 | 318 | 313
Percentage of Subjects | 0.6 [-0.6 to 1.9] | 45.6 [40.1 to 51.1] | 53.0 [47.5 to 58.6]

2. Secondary Outcome: Percentage of Subjects With an Investigator Rating of None or Mild on the 4-Grade FWS for Forehead Line Severity at Maximum Eyebrow Elevation
Description: The Investigator assessed the severity of the subject's forehead lines at maximum eyebrow elevation using the 4-grade FWS, where 0=none, 1=mild, 2=moderate, and 3=severe. The percentage of subjects with a score of "none" and "mild" are reported.
Time Frame: Day 30
Population: Intent-to-Treat: all randomized subjects with a score of "none" and "mild" on the FWS at maximum eyebrow elevation
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | Placebo (Normal Saline) Followed by OnabotulinumtoxinA Dose A | OnabotulinumtoxinA Dose B | OnabotulinumtoxinA Dose A
Number analyzed (Participants) | 156 | 318 | 313
Percentage of Subjects | 3.8 [0.8 to 6.9] | 90.3 [87.0 to 93.5] | 94.9 [92.4 to 97.3]

3. Secondary Outcome: Percentage of Subjects With ≥1-Grade Improvement From Baseline on the Investigator's FWS Rating of Forehead Line Severity at Rest
Description: The Investigator assessed the severity of the subject's forehead lines at rest using the 4-grade FWS, where 0=none, 1=mild, 2=moderate, and 3=severe. The percentage of subjects with at least a 1-grade improvement assessed by the Investigator are reported.
Time Frame: Baseline, Day 30
Population: Intent-to-Treat: all randomized subjects with at least a 1-grade improvement assessed by the Investigator on the FWS at rest
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | Placebo (Normal Saline) Followed by OnabotulinumtoxinA Dose A | OnabotulinumtoxinA Dose B | OnabotulinumtoxinA Dose A
Number analyzed (Participants) | 150 | 310 | 309
Percentage of Subjects | 18.7 [12.4 to 24.9] | 85.2 [81.2 to 89.1] | 84.8 [80.8 to 88.8]

4. Secondary Outcome: Percentage of Subjects Reporting Mostly Satisfied or Very Satisfied on the 5-Point Facial Line Satisfaction Questionnaire (FLSQ) Item 5
Description: The FLSQ consists of 13 questions that assess subject satisfaction and appearance-related impacts associated with facial lines. Item 5 on the FLSQ asks "How satisfied are you with the effect your treatment had on your facial lines?" Responses included: very satisfied, mostly satisfied, neither satisfied or dissatisfied, mostly dissatisfied, or very dissatisfied. The percentage of subjects reporting a score of mostly satisfied or very satisfied with treatment are reported.
Time Frame: Day 60
Population: Intent-to-Treat: all randomized subjects with data reported at this time point
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | Placebo (Normal Saline) Followed by OnabotulinumtoxinA Dose A | OnabotulinumtoxinA Dose B | OnabotulinumtoxinA Dose A
Number analyzed (Participants) | 155 | 317 | 313
Percentage of Subjects | 3.2 [0.4 to 6.0] | 81.4 [77.1 to 85.7] | 87.9 [84.2 to 91.5]

5. Secondary Outcome: Percentage of Subjects With ≥20-Point Improvement From Baseline on the Impact Domain of the FLSQ Among Subjects With Baseline Score ≥ 20 Points
Description: The FLSQ consists of 13 questions that assess subject satisfaction and appearance-related impacts associated with facial lines. The Impact Domain measures the subject's appearance-related and emotional impacts of treatment and is composed of 5 questions with a possible range of scores from 0 (worst) to 100 (best), using a transformed scale. Only subjects with baseline scores ≥ 20 are included in the analysis.
Time Frame: Baseline, Day 30
Population: Intent-to-Treat: all randomized subjects with baseline scores ≥ 20 on the Impact Domain of the FLSQ
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | Placebo (Normal Saline) Followed by OnabotulinumtoxinA Dose A | OnabotulinumtoxinA Dose B | OnabotulinumtoxinA Dose A
Number analyzed (Participants) | 152 | 310 | 301
Percentage of Subjects | 19.7 [13.4 to 26.1] | 61.0 [55.5 to 66.4] | 76.1 [71.3 to 80.9]

6. Secondary Outcome: Percentage of Subjects With a ≥3-Point Improvement From Baseline on Item 4 of the 11-Point Facial Line Outcomes (FLO-11) Questionnaire©
Description: The FLO-11 assess the subject's psychological and appearance-related impacts associated with facial lines. Item 4 is "I look older than my actual age because of my facial lines" with a range of possible scores from 0 = not at all to 10 = very much. Only subjects with baseline scores ≥ 3 are included in the analysis.
Time Frame: Baseline, Day 30
Population: Intent-to-Treat: all randomized subjects with baseline scores ≥ 3 on Item 4 of the FLO-11
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | Placebo (Normal Saline) Followed by OnabotulinumtoxinA Dose A | OnabotulinumtoxinA Dose B | OnabotulinumtoxinA Dose A
Number analyzed (Participants) | 141 | 285 | 288
Percentage of Subjects | 9.9 [5.0 to 14.9] | 66.7 [61.2 to 72.1] | 77.1 [72.2 to 81.9]

7. Secondary Outcome: Time to Retreatment Eligibility
Description: Time to retreatment eligibility is defined as the number of days from treatment cycle 1 injection to the return to an Investigator FWS rating of moderate or severe at maximum eyebrow elevation. The FWS is a 4-grade scale, where 0=none, 1=mild, 2=moderate, and 3=severe. Only subjects who achieved a ≥ 2-grade improvement on both the Investigator and subject FWS ratings at maximum eyebrow elevation on Day 30 are included in the analysis.
Time Frame: 12 Months
Population: Intent-to-Treat: all randomized subjects who achieved a ≥ 2-grade improvement on both the Investigator and subject FWS ratings at maximum eyebrow elevation
Measure: Median (Standard Deviation); unit: Days
Arm/Group | Placebo (Normal Saline) Followed by OnabotulinumtoxinA Dose A | OnabotulinumtoxinA Dose B | OnabotulinumtoxinA Dose A
Number analyzed (Participants) | 1 | 143 | 161
Days | 64.0 (NA) — One incidence; therefore, SD not applicable | 120.0 (46.4) | 126.0 (53.7)

ADVERSE EVENTS:
Description: The Safety Population includes all subjects who received at least 1 study treatment injection and was used to assess AEs and SAEs. Subjects randomized to receive placebo in Period 1 who subsequently received open-label onabotulinumtoxinA Dose A in Period 2 are included in the onabotulinumtoxinA Dose A group for the Safety analysis.
Arm/Group | Placebo (Normal Saline) Followed by OnabotulinumtoxinA Dose A | OnabotulinumtoxinA Dose B | OnabotulinumtoxinA Dose A
Serious Adverse Events (participants affected / at risk) | 2/156 | 7/318 | 16/746
Other Adverse Events (participants affected / at risk) | 21/156 | 90/318 | 198/746
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (Normal Saline) Followed by OnabotulinumtoxinA Dose A (N=156) | OnabotulinumtoxinA Dose B (N=318) | OnabotulinumtoxinA Dose A (N=746)
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Abscess (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 2
Meningitis viral (Infections and infestations) | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 2 | 0
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant melanoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neuritis (Nervous system disorders) | 0 | 0 | 1
Temporal lobe epilepsy (Nervous system disorders) | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0/140 | 0/278 | 2/284
Alcoholism (Psychiatric disorders) | 0 | 0 | 1
Tonsillectomy (Surgical and medical procedures) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Normal Saline) Followed by OnabotulinumtoxinA Dose A (N=156) | OnabotulinumtoxinA Dose B (N=318) | OnabotulinumtoxinA Dose A (N=746)
Injection site bruising (General disorders) | 5 | 26 | 47
Injection site haematoma (General disorders) | 3 | 16 | 34
Nasopharyngitis (Infections and infestations) | 5 | 18 | 48
Headache (Nervous system disorders) | 8 | 30 | 69

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.